CLINICAL TRIAL: NCT03846310
Title: A Phase 1/1b Study to Evaluate the Safety and Tolerability of Immunotherapy Combinations in Participants With Lung Cancer
Brief Title: A Study to Evaluate Immunotherapy Combinations in Participants With Lung Cancer
Acronym: ARC-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-4 (AB928CSP0004)
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer; Nonsquamous Nonsmall Cell Neoplasm of Lung; Sensitizing EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — zimberelimab; Carboplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Arm A (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period. The RDE of etrumadenant will be determined in this part with escalating doses of etrumadenant in combination with standard doses of carboplatin/pemetrexed chemotherapy regimen in participants with Non-Small Cell Lung Cancer.
  Interventions: Drug: Etrumadenant; Drug: Carboplatin; Drug: Pemetrexed
- Dose Escalation Arm B (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period. The RDE of etrumadenant will be determined in this part with escalating doses of etrumadenant in combination with standard doses of carboplatin/pemetrexed chemotherapy regimen and pembrolizumab in participants with Non-Small Cell Lung Cancer.
  Interventions: Drug: Etrumadenant; Drug: Carboplatin; Drug: Pemetrexed; Drug: Pembrolizumab
- Dose Expansion Arm 1 (Experimental): Zimberelimab will be administered in combination with standard carboplatin and pemetrexed chemotherapy regimen in participants with Non-Small Cell Lung Cancer harboring a sensitizing EGFR mutation.
  Interventions: Drug: Zimberelimab; Drug: Carboplatin; Drug: Pemetrexed
- Dose Expansion Arm 2 (Experimental): The etrumadenant at RDE determined from the dose escalation phase will be administered in combination with standard carboplatin and pemetrexed chemotherapy regimen and zimberelimab in participants with Non-Small Cell Lung Cancer harboring a sensitizing EGFR mutation.
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Etrumadenant — Etrumadenant is an A2aR and A2bR antagonist
  Other Names: AB928
  Arms: Dose Escalation Arm A; Dose Escalation Arm B; Dose Expansion Arm 2
Drug: Zimberelimab — Zimberelimab is a fully human anti-PD-1 monoclonal antibody
  Other Names: AB122
  Arms: Dose Expansion Arm 1; Dose Expansion Arm 2
Drug: Carboplatin — Carboplatin administered as part of standard chemotherapy regimen
Drug: Pemetrexed — Pemetrexed administered as part of standard chemotherapy regimen
Drug: Pembrolizumab — Pembrolizumab is a humanized anti-PD-1 monoclonal antibody
  Arms: Dose Escalation Arm B

SUMMARY:
This is a Phase 1/1b, multicenter, open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic, and clinical activity of etrumadenant (AB928) in combination with carboplatin and pemetrexed, with or without an anti-PD-1 antibody (pembrolizumab or zimberelimab), in participants with non-squamous Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
In the dose-escalation phase, escalating doses of etrumadenant in combination with carboplatin and pemetrexed at standard doses (Arm A), and etrumadenant in combination with carboplatin, pemetrexed and pembrolizumab (Arm B), may be assessed in participants with advanced NSCLC. Eligible participants will receive oral administration of etrumadenant as well as IV infused carboplatin, pemetrexed, with or without pembrolizumab in this phase. The recommended dose for expansion (RDE) of etrumadenant will be determined upon completion of the dose-escalation phase.

In the dose-expansion phase, zimberelimab in combination with carboplatin and pemetrexed (Arm 1), and etrumadenant at RDE in combination with carboplatin, pemetrexed, and zimberelimab (Arm 2) may be assessed in eligible NSCLC participants who harbor an EGFR mutation and have progressed on EGFR Tyrosine Kinase Inhibitor (TKI) treatment(s).

Overall duration of treatment will depend on how well the treatment is tolerated.

Treatment may continue until unacceptable toxicity or progressive disease or other reasons specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants; age ≥ 18 years
* Pathologically confirmed nonsquamous NSCLC that is metastatic, locally advanced, or recurrent with progression
* Arm A participants must fulfill one of the following:

  * Participant has a genetic alteration (mutation or rearrangement) and has received all available targeted therapy. Previous treatment with chemotherapy or PD-1/-L1 therapy is not allowed.
  * Participant has not received any therapy for the disease under study and standard therapy is refused.
  * Participant has progressed on PD-1/-L1 therapy (monotherapy or combination regimen). Previous treatment with chemotherapy is not allowed.
  * Participant has progressed on PD-1/-L1 therapy (monotherapy or combination regimen) and has received less than 4 cycles of carboplatin/pemetrexed and further chemotherapy is appropriate.
  * Participant has received any number of prior treatments and is without alternative or curative therapy.
* Arm B participants must fulfill one of the following:

  * Participant has a genetic alteration (mutation or rearrangement) and has received all available targeted therapy. Previous treatment with chemotherapy or PD-1/-L1 therapy is not allowed.
  * Participant has not received any therapy for the disease under study and standard therapy is refused.
  * Participant has received any number of prior treatments and is without alternative or curative therapy.
* Arm 1 and Arm 2 participants must have a sensitizing epidermal growth factor receptor (EGFR) mutation with disease progression or treatment intolerance after one or more approved TKIs. Previous treatment with chemotherapy or PD-1/L-1 therapy is not allowed.
* No TKI therapy within 5 days of Cycle 1 Day 1
* The last dose of previous investigational therapy is at least 4 weeks or 5 half-lives prior to Cycle 1 Day 1.
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Confirm that an archival tissue sample is available and ≤ 24 months old; if not, a new biopsy of a tumor lesion should be obtained at screening
* Adequate organ and marrow function

Exclusion Criteria:

* Use of any live vaccines against infectious diseases within 4 weeks (28 days) of initiation of investigational product
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 30 days after the last dose of etrumadenant, 90 days after the last dose of zimberelimab or pembrolizumab, or 6 months after the last dose of pemetrexed, whichever is longer
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer
* Prior use of an adenosine pathway targeting agent
* Due to potential for drug-drug interactions with etrumadenant, participants must not have had:

  * Treatment with breast cancer resistance protein substrates or P-glycoprotein with a narrow therapeutic window, administered orally within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
  * Treatment with known strong cytochrome P450 3A4 (CYP3A4) inducers and strong CYP3A4 inhibitors within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Events | From first study treatment administration until up to 90 days after the last dose (Approximately 1 year)
Percentage of participants who experience a Dose Limiting Toxicity | From first study treatment administration through Day 21

SECONDARY OUTCOMES:
Percentage of participants with anti-drug antibodies to zimberelimab | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 days post last dose (i.e. in total approximately 5 months).
Plasma concentration of etrumadenant | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 days post last dose (i.e. in total approximately 5 months).
Serum concentration of zimberelimab | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months) and 30 days post last dose (i.e. in total approximately 5 months).
Progression Free Survival (PFS) | From start of treatment up to the first occurrence of progressive disease or death from any cause, whichever occurs first (up to approximately 3-5 years)
Duration of Response | From the date of first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
Percentage of Participants with Disease Control (complete response, partial response, or stable disease) for >6 months | From study enrollment until disease progression or loss of clinical benefit (up to approximately 3-5 years)
Percentage of participants with Objective Response | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (up to approximately 3-5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (22):
- United States (8):
  - Arizona Cancer Research Center (ACRC), Tucson, Arizona
  - SCRI Florida Cancer Specialists - South, Fort Myers, Florida
  - SCRI Florida Cancer Specialists - North, Tavares, Florida
  - SCRI Tennessee Oncology - Nashville, Nashville, Tennessee
  - USO Texas Oncology - Dallas (Baylor Charles A. Sammons Cancer Center), Dallas, Texas
  - USO Virginia Cancer Specialist, Fairfax, Virginia
  - USO Virginia Oncology Associates, Norfolk, Virginia
  - Medical Oncology Associates/Summit Cancer Center, Spokane, Washington
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (7):
  - The Catholic University of Korea St. Vincent Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si
  - Bundang CHA Medical Center, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Centre, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Suwon
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy/

REFERENCES:
- See also: ARC-4 - Public website — https://trials.arcusbio.com/study/?id=ARC-4